CLINICAL TRIAL: NCT01484054
Title: Dispensing Evaluation of Lens Comfort and Subjective Vision of an Etafilcon A With Print and PVP Lens for Dark Eyes
Brief Title: Dispensing Evaluation of Subjective Comfort, Vision, and Handling of a New Lens Compared to a Marketed Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-005128
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Refractive Ametropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EAPVPDE/EADE (Other): etafilcon A with embedded print and PVP lens for dark eyes worn daily during the first period of 7-9 days, then etafilcon A control lens worn daily during the second period of 7-9 days, with 1-3 days of wash-out time between the 2 periods.
  Interventions: Device: etafilcon A with print and PVP for dark eyes (EAPVPDE); Device: etafilcon A control lens (EADE)
- EADE/EAPVPDE (Other): etafilcon A control lens worn daily during the first period of 7-9 days, then etafilcon A with embedded print and PVP for dark eyes lens worn daily during the second period of 7-9 days, with 1-3 days of wash-out time between the 2 periods.
  Interventions: Device: etafilcon A with print and PVP for dark eyes (EAPVPDE); Device: etafilcon A control lens (EADE)

INTERVENTIONS:
Device: etafilcon A with print and PVP for dark eyes (EAPVPDE) — A daily disposable contact lens
Device: etafilcon A control lens (EADE) — A marketed daily disposable contact lens

SUMMARY:
To evaluate and compare the performance of a new contact lens to a marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be a healthy adult at least 18 years of age and no more than 34 years of age.
* The subjects must be female, dark eye Caucasian, Non-Hispanic habitual soft contact lens wearer (both eyes).
* The subject rated the Concept Statement positively (i.e., a rating of 4 or 5). If not the subject is not eligible to participate.
* The subject must have no known ocular or systemic allergies that might interfere with contact lens wear.
* The subject must have no known systemic disease, or need for medication, which might interfere with contact lens wear.
* The subject's optimal vertexed spherical equivalent distance correction must be between-1.00 and -4.00D.
* Any cylinder power must be:<=0.75D.
* The subject must have visual acuity best correctable to 20/25 or better for each eye.
* The subject must have normal eyes (no ocular medications or ocular infection of any type).
* The subject must read and sign the Statement of Informed Consent.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear.
* Systemic disease, autoimmune disease, or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or worse) corneal edema, corneal neovascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Any color deficiencies (color blindness) - to the best of the subject's knowledge.
* Pregnancy or lactation.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Habitual contact lens type is toric, multifocal, or is worn as extended wear.
* Subject presents with one dark iris color and one light iris color
* Subject has heterochromia iridis (a difference in color between parts of one iris)
* The subject is an employee or family member of the clinical study site.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Bloomfield, Connecticut
  - Tallahassee, Florida
  - Overland Park, Kansas
  - Jamestown, New York
  - Kingston, Pennsylvania
  - Moon Township, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of those 103 enrolled subjects, 3 subjects did not receive the study article.
Groups:
- EAPVPDE/EADE: etafilcon A with embedded print and PVP for dark eyes lens worn daily during the first period of 7-9 days then etafilcon A control lens worn daily during the second period of 7-9 days with a 1-3 day of wash-out time between 2 periods.
- EADE/EAPVPDE: etafilcon A control lens worn daily during the first period of 7-9 days then etafilcon A with embedded print and PVP for dark eyes lens worn daily during the second period of 7-9 days with a 1-3 day of wash-out time between 2 periods.
Period: Period 1
Arm/Group | EAPVPDE/EADE | EADE/EAPVPDE
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | EAPVPDE/EADE | EADE/EAPVPDE
Started | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all enrolled subjects who received study lenses.
Groups:
- All Subjects: All enrolled subjects who received study lenses.
Arm/Group | All Subjects
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.07 (4.879)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Overall Quality of Lens Vision Using the Contact Lens User Evaluation (CLUE) Questionnaire
Description: The overall quality of lens vision was assessed using the CLUE questionnaire after 7-9 days of follow-up. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range from 0-120.
Time Frame: After 7 to 9 days of lens wear
Population: Analysis was conducted on subjects who successfully complete the study without a protocol deviation affecting at least one primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- EAPVPDE: A daily disposable contact lens.
- EADE: A marketed daily disposable contact lens
Arm/Group | EAPVPDE | EADE
Number analyzed (Participants) | 92 | 92
units on a scale | 54.06 (2.538) [48.56 to 59.57] | 53.06 (2.537) [47.56 to 58.57]
Statistical Analysis 1: Comparison: EAPVPDE vs EADE; The alternative hypothesis is that etafilcon A with PVP lenses is non-inferior to etafilcon A control lenses for the Overall Quality of Lens Vision at 7-9 days of follow-up; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -5 points(CLUE) was used; Mixed Models Analysis; Least square mean difference = 1.00, 95% CI 2-sided [-3.20 to 5.20], Standard Error of Mean 2.117

2. Primary Outcome: Subject Reported Overall Lens Comfort Using the Contact Lens User Evaluation (CLUE) Questionnaire
Description: The overall lens comfort was assessed using the CLUE questionnaire after 7-9 days of follow-up.The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: After 7 to 9 days of lens wear
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | EAPVPDE | EADE
Number analyzed (Participants) | 92 | 92
units on a scale | 53.61 (2.201) [49.27 to 57.95] | 48.91 (2.197) [44.58 to 53.25]
Statistical Analysis 1: Comparison: EAPVPDE vs EADE; The alternative hypothesis is that etafilcon A with PVP lenses is non-inferior to etafilcon A control lenses for the Overall Lens Comfort at 7-9 days of follow-up; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -5 points(CLUE) was used; Mixed Models Analysis; Least square mean difference = 4.70, 95% CI 2-sided [-0.79 to 10.19], Standard Error of Mean 2.772

3. Primary Outcome: Subject Reported Overall Lens Handling Using the Contact Lens User Evaluation (CLUE) Questionnaire
Description: The overall lens handling was assessed using the CLUE questionnaire after 7-9 days of follow-up. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: After 7 to 9 days of lens wear
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | EAPVPDE | EADE
Number analyzed (Participants) | 92 | 92
units on a scale | 61.21 (1.847) [57.56 to 64.86] | 51.77 (1.842) [48.12 to 55.41]
Statistical Analysis 1: Comparison: EAPVPDE vs EADE; Ho: The test lens is non-inferior to the active comparator lens for Handling at 7-9 days follow-up; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -5 points(CLUE) was used; Mixed Models Analysis; Least square mean difference = 9.44, 95% CI 2-sided [5.81 to 13.07], Standard Error of Mean 1.829

ADVERSE EVENTS:
Time Frame: Adverse events were recorded when the subjects were exposed to the Investigational lenses.
Groups:
- EAPVPDE: etafilcon A material incorporating PVP in the blister packaging solution.
- EADE: etafilcon a existing, daily disposable contact lens.
Arm/Group | EAPVPDE | EADE
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other